CLINICAL TRIAL: NCT06821282
Title: Surveillance of Antimicrobial Resistance in Semirural Kinshasa, Democratic Republic of Congo: a Feasibility Study
Brief Title: Surveillance of AMR in DRC
Acronym: SARKIN
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Kinshasa (Other); Mahidol University (Other); Institut National de Recherche Biomédicale (INRB). Kinshasa, Democratic Republic of Congo (Unknown); Department of Infectious Diseases, The Alfred Hospital and School of Translational Medicine, Monash University, Melbourne, Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: MID24001
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Bacteremia
Keywords: Antimicrobial resistance (AMR); Surveillance; Malaria; Africa; Democratic Republic of Congo
MeSH Terms: conditions — Bacteremia; Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study addresses knowledge gaps regarding antimicrobial resistance (AMR) in sub-Saharan Africa, focusing on evaluating the feasibility of AMR surveillance and enhancing local research capacity. Conducted at a general referral hospital in semirural Kinshasa, DRC, the study will investigate bacterial infections, their resistance profiles, and related risk factors, including co-infections such as malaria.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) is a significant global health threat, but its full impact in many African regions is still poorly understood. In collaboration with the Kinshasa School of Public Health, the Institut National de la Recherche Biomédicale (INRB) of DRC, and the University of Oxford, this study will assess the feasibility of implementing AMR surveillance in a general referral hospital in semirural Kinshasa, where onsite microbiological testing is currently unavailable. A key objective is to strengthen local research capacity by training staff in patient identification and specimen collection for AMR surveillance. The study will include patients over six months of age with suspected bloodstream infections at the time of hospital admission who agree to participate and from whom informed consent has been obtained. The focus is on community-acquired infections, excluding patients with significant prior healthcare or antibiotic exposure. Blood samples will be analyzed at INRB to determine the bacterial cause of infections, evaluate antimicrobial resistance levels, and identify associated risk factors, including co-infection with Plasmodium falciparum. Study results will be shared promptly with the hospital team to aid in patient management. Participants will be followed up for 28 days post-admission.

ELIGIBILITY:
Patients older than six months who present with a clinically suspected bloodstream infection upon admission to the hospital, or who have been hospitalized for less than 48 hours, and provide written consent (or consent from their caregiver/legal guardian) to participate will be included. Patients with a significant history of healthcare exposure and those with any contraindications for phlebotomy as determined by the clinician's judgment, will be excluded.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 6 months, admitted to the Hospital with a clinical suspicion of bloodstream infection.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment process | Duration of recruitment, about six months
  The feasibility of establishing AMR surveillance at a referral hospital in Kinshasa, DRC will be assessed by evaluating the number of eligible patients, the number of patients who consent and the number of enrolled patients by syndrome each month with blood samples collected.
Intervention delivery | Duration of recruitment, about six months
  Another key feasibility metric will be to assess the proportion of samples with final results from the microbiology lab, the proportion of possibly contaminated blood cultures, and the proportion of positive cultures with antimicrobial susceptibility testing.
Processing time | Duration of recruitment, about six months
  The time from patient enrolment to blood sample collection and to transfer to the laboratory will be measured.
Number of Bacterial Bloodstream Infections | Duration of recruitment, about 6 months
  The characterization of bacterial bloodstream infections (BSI) will be assessed by the frequency of positive blood cultures in patients with suspected BSI, the proportion of severe falciparum malaria patients diagnosed with concomitant BSI, and the outcome of BSI, in-hospital mortality, and 28-day mortality.
Antimicrobial Susceptibility | Duration of recruitment, about six months
  Antimicrobial resistance patterns of bacterial isolates.
Co-infection | Duration of recruitment, about six months
  Proportion of severe falciparum malaria patients diagnosed with concomitant BSI.
Outcome | Study duration, plus 4 weeks
  In-hospital and 28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Fanello, Dr., Principal Investigator — Centre for Tropical Medicine and Global Health, Nuffield Department of Medicine, University of Oxford, United Kingdom (UK); Sue J Lee, Dr., Principal Investigator — Mahidol-Oxford Research Unit (MORU), Faculty of Tropical Medicine, Mahidol University, Bangkok,Thailand
Locations (1):
- Kinshasa, Democratic Republic of Congo, Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Key variables on pathogen identified and AMR will be shared through GRAM (URL: https://www.tropicalmedicine.ox.ac.uk/gram) All other data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of activities and reporting
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing